CLINICAL TRIAL: NCT04455776
Title: Incidence of Adverse Events During Propofol Sedation for Magnetic Resonance Imaging in Pediatric Patients
Brief Title: Safety Evaluation of Propofol Sedation for Magnetic Resonance Imaging in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Denis SCHMARTZ, Head of Anesthesiology department, Brugmann University Hospital
Other Study IDs: CHUB_PEDIRM
Record Dates: First submitted 2020-06-25; First posted 2020-07-02 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Multiparametric Magnetic Resonance Imaging; Propofol Adverse Reaction; Sedation Complication; Anesthesia; Adverse Effect
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Propofol — Sedation by propofol

SUMMARY:
Propofol is often used for sedation in children undergoing magnetic resonance imaging. The investigators will perform a chart review of 4 month of activity (about 100 cases) and review the incidence and severity of adverse events of this sedation technique.

DETAILED DESCRIPTION:
Magnetic resonance imaging in children, especially under 6 years of age, is often performed under sedation. Propofol is a common drug used in this settings. In our institution, sedation is most often done by a propofol bolus of 2-5 mg/kg in order to reach a deep level of sedation as defined by Coté et al. If judged necessary by the attending anaesthesiologist, a additional propofol bolus of 0.5-1 mg/kg may be given. For longer lasting exams, the attending anaesthesiologist can chose to use a continuous infusion of propofol. The investigators will review the charts of 4 month of magnetic resonance imaging, which will give us a cohort of about 100 patients. Baseline characteristics, detailed sedation technique used will be recorded. Adverse events defined as:

* Oxygen desaturation measured by transcutaneous oximetry SpO2≤94%
* hypercapnia measure by end-tidal CO2 >45 mm Hg
* movement of the patient

Assuming a non-normal distribution (tested by a Kolmogorov-Smirnov test), variables will be reported as median and interquartile range. Statistical tests will be done by non-parametric tests, Mann Whitney U. Non continuous variables will be analyzed by a Chi-square test.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients scheduled for MRI under sedation by an anaesthesiologist
* Age < 16 years

Exclusion Criteria:

* Age > 16 years
* Sedation performed by a non-anesthesiologist

Max Age: 16 Years | Sex: All
Age Groups: Child
Study Population: Pediatric patients under 16 years undergoing magnetic resonance imaging under propofol sedation.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2020-07-03 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Hypoxemia | 90 minutes
  Arterial desaturation defined as number of episodes with an SpO2≤94%
Hypercapnia | 90 minutes
  Hypercapnia, defined as number of episodes with an ETCO2 > 45 mm HG
Movements | 90 minutes
  Number of patient movements interfering with the MRI exam

CONTACTS AND LOCATIONS:
Overall Officials: Denis Schmartz, MD, Principal Investigator — CHU Brugmann
Locations (1):
- Hôpital Universitaire des Enfants Reine Fabiola, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No